CLINICAL TRIAL: NCT03014570
Title: Testing the Implementation of EIT-4-BPSD
Acronym: EIT-4_BPSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Barbara Resnick, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00069354
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Dementia; Behavioral and Psychological Symptoms of Dementia (BPSD)
Keywords: behavior,; apathy; mood; function; cognition
MeSH Terms: conditions — Dementia; Behavior; Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education-Only Control (Active Comparator): This arm includes the education provided to all sites (this is Step 2 of the EIT-4-BPSD intervention). The sites are given the opportunity to decide how they want the education around management of behavioral symptoms to occur-face-to-face by a research staff member, via a powerpoint they can use on their own or via a webinar.
  Interventions: Behavioral: Education-only Control
- EIT-4-BPSD (Experimental): This arm includes the four step intervention: 1. Assessment of the environment and policies; 2. Education of staff; 3. Establishing person-centered care plans; and 4. Mentoring and motivating staff. We provide the sites with a research nurse who works with an identified stakeholder group and champion within the facility and visits the settings monthly, connects by email weekly to complete the four intervention steps. The implementation process is guided by the Evidence Integration Triangle (EIT) framework. The EIT brings together evidence and key stakeholders from the facility to influence care practices. EIT includes: participatory implementation processes, provision of practical evidence-based interventions, and pragmatic measures of progress toward goals.
  Interventions: Behavioral: EIT-4-BPSD

INTERVENTIONS:
Behavioral: EIT-4-BPSD — This arm includes the four step intervention: 1. Assessment of the environment and policies; 2. Education of staff; 3. Establishing person-centered care plans; and 4. Mentoring and motivating staff. We provide the sites with a research nurse who works with an identified stakeholder group and champion within the facility and visits the settings monthly, connects by email weekly to complete the four intervention steps. The implementation process is guided by the Evidence Integration Triangle (EIT) framework. The EIT brings together evidence and key stakeholders from the facility to influence care practices. EIT includes: participatory implementation processes, provision of practical evidence-based interventions, and pragmatic measures of progress toward goals.
  Arms: EIT-4-BPSD
Behavioral: Education-only Control — This arm includes step 2 only of the EIT-4-BPSD. Facilities are provided with education abouthow to provide behavioral interventions for behavioral symptoms associated with dementia. They can have the education face-to-face or via a powerpoint or webinar.
  Arms: Education-Only Control

SUMMARY:
This pragmatic trial focuses on implementation of an evidence based process to increase person-centered management of behavioral and psychological symptoms of dementia (BPSD) in nursing homes, referred to as EIT-4-BPSD. The findings from this study will add to what is known about implementation of effective interventions in nursing homes, will serve as a model for other programs and care approaches, and will help facilities and staff implement quality person-centered care, which is the goal of the National Partnership to Improve Dementia Care and Reduce Antipsychotic Use in Nursing Homes.

DETAILED DESCRIPTION:
Behavioral and Psychological Symptoms of Dementia (BPSD) include aggression, agitation, depression, anxiety, apathy and hallucinations and are exhibited by up to 90% of nursing facility residents with dementia. BPSD result in negative health outcomes decline in physical functioning and high cost of care. In addition, BPSD put residents at risk for inappropriate use of antipsychotic drugs and other restraining methods that reduce function, increase social isolation, and increase risk of physical abuse. Prior NIH-funded clinical trials show that behavioral approaches reduce BPSD. These behavioral approaches are endorsed as the first line of treatment for BPSD. In fact, the Centers for Medicare and Medicaid Services (CMS) National Partnership to Improve Dementia Care and Reduce Antipsychotic Use in Nursing Homes requires that care for residents with dementia be delivered using person-centered behavioral approaches. Despite regulatory requirements, less than 2% of nursing homes (also referred to as facilities) consistently implement these approaches. Established barriers to use of behavioral approaches include limited knowledge, skills, and experience with non-pharmacological approaches, beliefs in the superiority of psychotropic medications over behavioral interventions, and lack of staff motivation to use non-pharmacologic strategies consistently. The proposed project responds to this gap between knowledge and practice. A novel implementation approach will be tested to assure that staff in nursing homes [i.e., those who provide direct care to residents] use non-pharmacologic, behavioral approaches for the management of BPSD.

To advance the CMS National Partnership, a comprehensive compendium of peer-reviewed/expert-endorsed resources was developed for utilizing person-centered, behavioral approaches for BPSD (the Nursing Home Toolkit: www.nursinghometoolkit.com). The Toolkit has resources that support a theoretically-based 4-step approach that we found effective in prior implementation work. The four steps include: 1. Assessment of the environment and policies; 2. Education of staff; 3. Establishing person-centered care plans; and 4. Mentoring and motivating staff. While the Toolkit is free and accessible, staff in nursing homes need help with implementation. Implementation of the theoretically based 4-step approach is guided by the Evidence Integration Triangle (EIT) framework. The EIT brings together evidence and key stakeholders from the facility to influence care practices. EIT includes: participatory implementation processes, provision of practical evidence-based interventions, and pragmatic measures of progress toward goals. This implementation framework was merged with the 4-step approach and the Nursing Home Toolkit resources to develop the intervention, EIT-4-BPSD. The goal is to demonstrate that EIT-4-BPSD is an implementation strategy that enables staff in nursing homes to reduce BPSD using behavioral approaches while optimizing function, preventing adverse events and improving quality of life of residents. A Hybrid III cluster randomized trial will be done with 50 nursing facilities randomized to EIT-4-BPSD or Education Only (EO). The aims are:

Primary Aim 1: To implement and test the implementation of EIT-4-BPSD. Facility Level Outcome: Research question: Do facilities exposed to EIT-4-BPSD demonstrate evidence of implementation at 12 months evaluated by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) criteria? For evaluation of Effectiveness within RE-AIM: Resident Level Outcomes: Hypothesis: Residents in EIT-4-BPSD facilities will experience less BPSD, maintain or improve function, have reduced use of psychotropic medications, experience fewer adverse events, and have improved quality of life compared to residents in EO facilities. We will measure these outcomes at baseline, 4 and 12 months post implementation of the intervention. Facility Level Outcomes: Hypotheses: (1) EIT-4-BPSD facilities will demonstrate improvements in Environment and Policy assessments that reflect support for behavioral approaches for BPSD, and will have a greater percentage of residents with behavioral approaches incorporated into their care plans at 12 months post-implementation when compared to EO facilities; (2) We will examine Maintenance of EIT-4-BPSD facility outcomes at 12 months and then at 24 months post-implementation.

Primary Aim 2: Evaluation of the Feasibility, Utility and Cost of EIT Approach in EIT-4-BPSD Facilities. Using descriptive and qualitative data captured during the intervention and from focus groups at 12 months,use of the EIT strategy and the participatory implementation process with the Stakeholder Team and facility staff will be evaluated. In addition a description of the costs of implementation using an activity-based costing method will be completed.

This study will add critical knowledge to what little is known about implementation of effective interventions in nursing facilities. It will serve as an implementation model with potential to be widely disseminated. In addition, the study will demonstrate how facilities can implement person-centered dementia care and decrease BPSD, the ultimate goal of the CMS National Partnership.

ELIGIBILITY:
Inclusion Criteria:

Living in the nursing home; 55 years of age or older; score 0-12 on the Brief Interview of Mental Status

Exclusion Criteria:

* Enrolled in hospice
* in the nursing home for short stay rehabilitation

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2016-04; Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Behrens L, Boltz M, Riley K, Eshraghi K, Resnick B, Galik E, Ellis J, Kolanowski A, Van Haitsma K. Process evaluation of an implementation study in dementia care (EIT-4-BPSD): stakeholder perspectives. BMC Health Serv Res. 2021 Sep 23;21(1):1006. doi: 10.1186/s12913-021-07001-2. PMID 34551782
- [Derived] Kolanowski A, Zhu S, Van Haitsma K, Resnick B, Boltz M, Galik E, Behrens L, Eshraghi K, Ellis J. 12-month trajectory and predictors of affect balance in nursing home residents living with dementia. Aging Ment Health. 2022 Aug;26(8):1686-1692. doi: 10.1080/13607863.2021.1947964. Epub 2021 Jul 12. PMID 34253099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 553 residents enrolled into the study from 55 care communities from Maryland and Pennsylvania .
Pre-assignment Details: there were no significant events prior to the implementation of the study. No one was excluded.
Groups:
- Education-Only Control: This arm includes the education provided to all sites (this is Step 2 of the EIT-4-BPSD intervention).
  Education-only Control: This arm includes step 2 only of the EIT-4-BPSD. Facilities are provided with education abouthow to provide behavioral interventions for behavioral symptoms associated with dementia. They can have the education face-to-face or via a powerpoint or webinar.
  There were 27 sites randomized to control which included 248 participants.
- EIT-4-BPSD: This arm includes the four step intervention: 1. Assessment of the environment and policies; 2. Education of staff; 3. Establishing person-centered care plans; and 4. Mentoring and motivating staff. We provide the sites with a research nurse who works with an identified stakeholder group and champion within the facility and visits the settings monthly, connects by email weekly to complete the four intervention steps. The implementation process is guided by the Evidence Integration Triangle (EIT) framework. The EIT brings together evidence and key stakeholders from the facility to influence care practices. EIT includes: participatory implementation processes, provision of practical evidence-based interventions, and pragmatic measures of progress toward goals.
  There were 28 sites randomized to treatment which included 305 participants.
Period: Overall Study
Arm/Group | Education-Only Control | EIT-4-BPSD
Started | 248 (All of the intervention activities have been completed the date of completion was March 2020) | 305 (all of the intervention activities have been completed. the date of completion was march 2020)
Completed | 123 (All intervention activities were completed March 2020.) | 174 (all intervention activities were completed march 2020)
Not Completed | 125 | 131
Not completed — COVID-19 Restrictions | 38 | 24
Not completed — Death | 70 | 79
Not completed — Transfer from facility | 11 | 14
Not completed — Hospitalized | 5 | 3
Not completed — Transfer within facility | 1 | 0
Not completed — Site refusal | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education-Only Control | EIT-4-BPSD | Total
Number analyzed (Participants) | 248 | 305 | 553
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 248 | 305 | 553
Age, Continuous [Mean (Standard Deviation); unit: years of age] | 84 (10) | 82 (7) | 83 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 225 | 398
  Male | 75 | 80 | 155
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 83 | 134
  White | 197 | 222 | 419
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 248 | 305 | 553

OUTCOME MEASURES:

1. Primary Outcome: Physical Function as Determined by Barthel Index
Description: The Barthel index has a score range of 0-100 with higher scores indicating higher physical function
Time Frame: Baseline, 4 months and 12 months
Population: Older adults in nursing analysis was a repeated measures
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education-Only Control | EIT-4-BPSD
Number analyzed (Participants) | 123 | 174
score on a scale
  12 months | 35.82 (27.75) | 31.36 (26.88)
  4 months | 33.63 (30.33) | 33.93 (28.06)
  Baseline | 36.52 (30.72) | 36.56 (29.82)

2. Primary Outcome: Depression as Determined by the Cornell Scale for Depression in Dementia
Description: The Cornell scale ranges from 0-19 with higher scores representing more depressive symptoms
Time Frame: Baseline, 4 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education-Only Control | EIT-4-BPSD
Number analyzed (Participants) | 123 | 174
score on a scale
  12 months | 1.72 (2.5) | 1.86 (3.12)
  4 months | 3.91 (4.58) | 3.81 (4.15)
  Baseline | 4.11 (4.57) | 4.39 (3.81)

3. Primary Outcome: Agitation as Assessed by the Cohen-Mansfield Agitation Inventory (CMAI)
Description: The CMAI score ranges from 0-70 with higher scores indicating more agitation
Time Frame: Baseline, 4 months, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- EIT-4-BPSD: This arm includes the four step intervention: 1. Assessment of the environment and policies; 2. Education of staff; 3. Establishing person-centered care plans; and 4. Mentoring and motivating staff. We provide the sites with a research nurse who works with an identified stakeholder group and champion within the facility and visits the settings monthly, connects by email weekly to complete the four intervention steps.
  EIT-4-BPSD: This arm includes the four step intervention: 1. Assessment of the environment and policies; 2. Education of staff; 3. Establishing person-centered care plans; and 4. Mentoring and motivating staff. We provide the sites with a research nurse who works with an identified stakeholder group and champion within the facility and visits the settings monthly, connects by email weekly to complete the four intervention steps.
Arm/Group | Education-Only Control | EIT-4-BPSD
Number analyzed (Participants) | 123 | 174
score on a scale
  12 months | 20.42 (7.73) | 19.68 (6.92)
  4 months | 20.54 (7.74) | 20.24 (7.46)
  Baseline | 20.66 (8.34) | 21.32 (8.38)

ADVERSE EVENTS:
Time Frame: Over 12 months
Description: There were no adverse events.
Arm/Group | Education-Only Control | EIT-4-BPSD
All-Cause Mortality (participants affected / at risk) | 70/248 | 79/305
Serious Adverse Events (participants affected / at risk) | 0/248 | 0/305
Other Adverse Events (participants affected / at risk) | 0/248 | 0/305

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT03014570/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03014570/ICF_001.pdf